CLINICAL TRIAL: NCT05660668
Title: Comparative Assessment of Failure Rate of Fixed Lingual Retainer in Finished Orthodontic Cases Between Two Types of Light Cured Resin Composite. A Randomized Clinical Trial
Brief Title: Comparative Assessment of Failure Rate of Fixed Lingual Retainer Between Two Types of Light Cured Resin Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Saied, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORTHO 3-3-3
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Orthodontic Retainer
MeSH Terms: interventions — Transbond LR; Transbond XT

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbond LR (Experimental): in finished orthodontic cases a light cured resin composite (Transbond LR) will be added on fixed lingual retainer to see the failure rate (detachment) with follow up every month for 6 months
  Interventions: Other: Transbond LR
- Transbond XT (Active Comparator): in finished orthodontic cases a light cured resin composite (Transbond XT) will be added on fixed lingual retainer to see the failure rate (detachment) with follow up every month for 6 months
  Interventions: Other: Transbond XT

INTERVENTIONS:
Other: Transbond LR — cleaning the lingual surface using oil free pumice then apply acid etch 35% phosphoric acid for 20 second then rinse then Transbond LR will be applied directly on the fixed retainer and lingual surface of the teeth then light cured.
  Other Names: 3m brand
  Arms: Transbond LR
Other: Transbond XT — cleaning the lingual surface using oil free pumice then apply acid etch 35% phosphoric acid for 20 second then rinse then Transbond XT will be applied directly on the fixed retainer and lingual surface of the teeth then light cured.
  Other Names: 3m brand
  Arms: Transbond XT

SUMMARY:
The study will be performed on human subjects with finished orthodontic treatment to see the failure rate(detachment) of fixed lingual retainer between two types of light cure resin composite

DETAILED DESCRIPTION:
The study consists of two groups, the intervention involve performing bonding of fixed lingual retainer with light cured composite Transbond LR which is manufactured specific for the fixed lingual retainer while the control group involve bonding of fixed lingual retainer by light cured composite Transbond XT with follow up every month for 6 month to see the failure rate(detachment) between the two types of composite

ELIGIBILITY:
Inclusion Criteria:

* Patient at the end of an orthodontic treatment requiring the subsequent application of a lingual and palatal fixed retainer
* good oral hygiene
* medically free

Exclusion Criteria:

* Facial trauma
* onychophagia
* habit of biting pencils or pens
* tooth mobility

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Failure rate( detachment rate) of fixed lingual retainer | the patient will be inspected after applying the fixed retainer every month for 6 months
  measured by inspection of any detachment partial or complete of the fixed lingual retainer

CONTACTS AND LOCATIONS:
Overall Officials: Fady Hussein, Assoc. prof, Study Director — Cairo unversity
Locations (1):
- Cairo unversity ,Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No